CLINICAL TRIAL: NCT02732873
Title: A Multicentre Study Evaluating the Treatment of Meniscal Defects With a Meniscal Repair Scaffold, FibroFix™ Meniscus
Brief Title: Porous Tissue Regenerative Silk Scaffold for Human Meniscal Cartilage Repair
Acronym: REKREATE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant not received - study not started
Sponsor: Orthox Limited (Industry)
Collaborators: Southmead Hospital, Bristol, UK (Unknown); Magdeburg University Hospital, Germany (Unknown); Brandenburg University Hospital, Germany (Unknown); BundeswehrKrankenhaus Ulm, Germany (Unknown); Universitat Autonoma de Barcelona (Other); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORX/2016/FM02
Record Dates: First submitted 2016-03-09; First posted 2016-04-11 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Repair of Meniscal Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FibroFix (Experimental)
  Interventions: Device: FibroFix Meniscal Scaffold

INTERVENTIONS:
Device: FibroFix Meniscal Scaffold — FibroFix™ Meniscus scaffold is a silk derived product developed to functionally replace the excised unstable meniscus following a meniscal tear.

SUMMARY:
The REKREATE project will be an international, multi-centre, non-randomised, prospective single-arm pivotal study. All study patients will receive the FibroFix™ Meniscus scaffold following the provision of informed consent. A study period of 1 year and extended follow up period of up to 3 years is planned , to enable a thorough and complete assessment of the performance of the device when implanted to replace removed or damaged meniscal tissue in humans. The test article for this multi-centre study is the FibroFix™ Meniscus scaffold, which has been developed for repair of defects of the meniscus.

ELIGIBILITY:
Inclusion Criteria:

* The subject (or guardian, if appropriate) has signed and dated a specific informed consent form;
* The subject is over the age of 18 and ≤55 years of age;
* The subject is able to comply with the protocol-defined pre-operative procedures, the post-operative clinical and radiographic evaluations and the recommended rehabilitation regimen as determined by the Investigator;
* The subject has a diagnosis of an MRI or arthroscopically confirmed irreparable medial meniscus defect;
* The meniscal defect should represent 25% or more of the meniscus and be amenable to implantation;
* The peripheral meniscal rim must be present;
* The subject has a functionally intact ACL (Anterior Cruciate Ligament);
* Haemoglobin >9g/dL and platelet count >100,000/mm3 prior to Day 1;
* No contraindication to general anaesthetic;
* Female subjects of child-bearing potential: a negative urine pregnancy test.

Exclusion Criteria:

* Subject is >55 years of age;
* The subject has a functionally deficient ACL;
* The subject has concomitant posterior cruciate ligament insufficiency of the involved knee or a concomitant injury that interferes with the subject's ability to comply with the recommended rehabilitation programme;
* The subject has a diagnosis of Grade IV Outerbridge Scale degenerative cartilage disease in the involved knee joint;
* Patients demonstrating an active local or systemic infection;
* Any condition, which in the judgment of the Investigator would preclude adequate evaluation of the FibroFix™ Meniscus scaffold and clinical outcome;
* The subject has a history of confirmed anaphylactoid reaction;
* The subject has received local administration of any type of corticosteroid or systemic administration of antineoplastic, immunostimulating, or immunosuppressive agents within 180 days prior to the scheduled surgery;
* The subject has evidence of osteonecrosis of the involved knee;
* The subject has a medical history that includes a confirmed diagnosis of rheumatoid or inflammatory arthritis, or relapsing polychondritis;
* If female and of child-bearing potential: evidence of a positive pregnancy test or a stated intention to become pregnant in the next 6-12 months;
* Current or recent (<3 months) participation in another device or drug study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Performance analysis of meniscal scaffold | At 12 months follow up
  Performance will be assessed by means of recognised, validated, standardised questionnaires (IKDC, Lysholm, Tegner)

SECONDARY OUTCOMES:
Clinical criteria: quality of life | At 12 months follow up
  Subjective assessments using internationally validated questionnaires EQ5D
Assessment of safety of meniscal scaffold - Incidence and severity of Adverse Events; incidence and severity of surgical complications | At 12 months follow up
  Incidence and severity of Adverse Events; incidence and severity of surgical complications
Clinical criteria: pain | At 12 months follow up
  At 12 months follow up